CLINICAL TRIAL: NCT02937532
Title: Effects of Combining Cognitive Behavioural Therapy With Task-oriented Balance Training for Reducing Fear of Falling in People With Chronic Stroke: A Randomized Controlled Trial
Brief Title: Fear of Falling in Patients With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shamay Ng, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SM_Ng
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Stroke
Keywords: Fear of falling; Fear avoidance behavior; cognitive behavioral therapy; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GHE + TOBT training (Placebo Comparator): Subjects will receive general health education and task-oriented balance training.
  Interventions: Behavioral: GHE + TOBT training
- CBT + TOBT training (Active Comparator): Subjects will receive group-based cognitive behavioral therapy and task-oriented balance training.
  Interventions: Behavioral: CBT + TOBT training

INTERVENTIONS:
Behavioral: GHE + TOBT training — All subjects will receive 45 minutes of GHE, followed by 45 minutes of TOBT program twice a week for 8 weeks.
  Arms: GHE + TOBT training
Behavioral: CBT + TOBT training — All subjects will receive 45 minutes of CBT, followed by 45 minutes of TOBT program twice a week for 8 weeks.
  Arms: CBT + TOBT training

SUMMARY:
The aim of the study is to evaluate whether combining cognitive-behavioral therapy (CBT) with task-oriented balance training (TOBT) is more effective than general health education (GHE) together with TOBT in promoting fear of falling and reducing activity avoidance behavior.

DETAILED DESCRIPTION:
The null hypothesis of this study will be that no significant difference in the efficacy of the two treatments (CBT + TOBT; GHE + TOBT) in promoting fear of falling and reducing fear avoidance behavior, and thus no significant difference in improving balance ability, reducing fall risks, improving health-related quality of life and community reintegration of people with stroke.

ELIGIBILITY:
Inclusion criteria: Subjects will be included if they

* are between 55 and 85 years of age;
* have been diagnosed with a first unilateral ischemic brain injury or intracerebral hemorrhage by magnetic resonance imaging or computed tomography within the previous 1 to 6 years;
* have been discharged from all rehabilitation services at least 6 months before program begins;
* are able to work independently at least 10 meters with or without an assistive device;
* have low balance self-efficacy (The Activities-specific Balance Confidence scale score of <80);
* are able to score > 7 out of 10 on the Chinese version of Abbreviated Mental Test; and
* are able to follow instructions and provide written informed consent.

Exclusion criteria: Subjects will be excluded if they

* have any additional medical, cardiovascular, orthopaedic, or psychiatric or psychological condition that would hinder proper treatment or assessment;
* have receptive dysphasia;
* have significant lower peripheral neuropathy; or
* are involved in a drug studies or other clinical trial.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
The Chinese version of the Activities-specific Balance Confidence scale (ABC-C) | 2 years
  The ABC-C be used to assess the level of fear of falling. The ABC-C consisted of 16 items reflecting the level of balance confidence from 0% (no confidence) to 100% (complete confidence)

SECONDARY OUTCOMES:
The Chinese version of the Lawton Instrumental Activities of Daily Living scale (IADL-C) | 2 years
  The IADL-C will be used to assess the ability of participants to live independently at home and community. The IADL-C included 9 items rating on a 3-point scale ranging from 0 to 18. Higher score indicates better performance.
The Chinese version of the Community Integration Measure (CIM-C) | 2 years
  The CIM-C consisted of 10 items soliciting on a 5-point scale in which the higher the score indicating the higher level of community integration.
The Chinese version of the Short Form General Health Questionnaire (SF-36-C) | 2 years
  The SF-36-C will be used to measure the health-related quality of life. It consisted of 2 scales, the physical health summary and mental health summary, rating on a two- to six-point Likert scale ranging from 0 to 100 each subscale. The higher the score indicating the higher level of health-related quality of life.
The Chinese version of the Survey of Activities and Fear of Falling in the Elderly (SAFFE-C) | 2 years
  The SAFFE-C will be used to assessed the level of fear avoidance behavior. It consisted of 22 items rating on a 4-point Likert scale ranging from 0 to 66. Lower score indicates less fear avoidance behaviors.
Berg Balance Scale | 2 years
  The BBS to assess the clinical balance. It consisted of 14 items with scoring from 0 to 56. The higher the score indicates the better balance performance.
The Short-form Physiological Profile Assessment (S-PPA) | 2 years
  The S-PPA will be used to assess the fall risk ranging from -2 to 4. The higher the score represents the lower the fall risk.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - The Hong Kong Polytechnic University, Hong Kong
  - The Hong Kong Polytechnic University, Hung Hom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu TW, Ng GYF, Chung RCK, Ng SSM. Decreasing Fear of Falling in Chronic Stroke Survivors Through Cognitive Behavior Therapy and Task-Oriented Training. Stroke. 2019 Jan;50(1):148-154. doi: 10.1161/STROKEAHA.118.022406. Epub 2018 Dec 7. PMID 30580723
- [Derived] Liu TW, Ng GYF, Ng SSM. Effectiveness of a combination of cognitive behavioral therapy and task-oriented balance training in reducing the fear of falling in patients with chronic stroke: study protocol for a randomized controlled trial. Trials. 2018 Mar 7;19(1):168. doi: 10.1186/s13063-018-2549-z. PMID 29514677